CLINICAL TRIAL: NCT05592340
Title: Impact of Restaurant Menu Carbon Footprint Labeling on Consumers Purchase Intentions and Perceptions
Brief Title: Restaurant Menu Carbon Footprint Labeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Christina Roberto, PHD, Mitchell J. Blutt and Margo Krody Blutt Presidential Associate Professor of Health Policy, Perelman School of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 849162
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Food Preferences
Keywords: food labeling; carbon footprint; dietary sustainability; eating; choice behavior
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to see a restaurant menu with one of two labeling schemes: 1) Control: calorie labels only; 2) Carbon footprint labels in addition to calorie labels. Participants will be instructed to select an entree to hypothetically order from the online restaurant menu. We will record participants' selections and match these to nutrition and carbon footprint information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Calorie labels shown on online restaurant menu
  Interventions: Behavioral: Exposure to calorie information
- Carbon footprint labels (Experimental): Carbon footprint labels shown on online restaurant menu next to every item in addition to calorie labels
  Interventions: Behavioral: Exposure to calorie information; Behavioral: Exposure to carbon footprint information

INTERVENTIONS:
Behavioral: Exposure to calorie information — Calories for all foods and beverages
Behavioral: Exposure to carbon footprint information — Carbon footprint labels for all foods and beverages
  Arms: Carbon footprint labels

SUMMARY:
This online randomized clinical trial will test the effects of restaurant menu carbon footprint labels on consumers' choices and perceptions of restaurant menu items.

DETAILED DESCRIPTION:
This online randomized clinical trial will test the effects of restaurant menu carbon footprint labels on consumers' choices and perceptions of restaurant menu items. Participants will be randomized to see a restaurant menu with one of two labeling schemes: 1) Control: calorie labels only; 2) Carbon footprint labels in addition to calorie labels. Participants will be instructed to select an entree to hypothetically order from an online restaurant menu. After selecting, they will be asked to answer questions about their perceptions of menu items and carbon footprint labels.The primary outcome will be the average carbon footprint of menu items chosen from the online menu.

ELIGIBILITY:
Inclusion Criteria:

* US adults aged 18 or older

Exclusion Criteria:

* Younger than 18
* Non-US

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2389 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Carbon footprint of selected menu item | The survey will take up to 20 minutes.
  Participants will select a menu item to purchase from the online restaurant menu. Outcome is carbon footprint of selected item.

SECONDARY OUTCOMES:
Calories in selected menu item | The survey will take up to 20 minutes.
  Participants will select a menu item to purchase from the online restaurant menu. Outcome is calorie content of selected item.
Perceived enjoyment of high-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all (1) to a great deal (5)
Perceived enjoyment of low-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all (1) to a great deal (5)
Perceived likelihood to order high-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all likely (1) to extremely likely (5)
Perceived likelihood to order low-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all likely (1) to extremely likely (5)
Perceived healthfulness of high-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all healthy (1) to extremely healthy (5)
Perceived healthfulness of low-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all healthy (1) to extremely healthy (5)
Estimated calories in high-carbon-footprint menu item | The survey will take up to 20 minutes.
  Open response variable
Estimated calories in low-carbon-footprint menu item | The survey will take up to 20 minutes.
  Open response variable
Perceived carbon footprint of high-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured with three multiple choice options: larger, smaller, or about the same carbon footprint compared to the typical menu item's carbon footprint
Perceived carbon footprint of low-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured with three multiple choice options: larger, smaller, or about the same carbon footprint compared to the typical menu item's carbon footprint
Perceived lowering of carbon footprint for high-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all (1) to a great deal (5)
Perceived lowering of carbon footprint for low-carbon-footprint menu item | The survey will take up to 20 minutes.
  This variable will be measured on a 5-point Likert scale ranging from not at all (1) to a great deal (5)
Noticing carbon footprint labels | The survey will take up to 20 minutes.
  Participants will respond "yes," "no," or "I don't know" to the item: "Think back to the beginning of this survey. When you were looking at the Just Salad menu, did you notice any labels (other than calorie information or price) next to or beneath the food items?"
Label influence | The survey will take up to 20 minutes.
  If participants responded "yes" to noticing labels, they will respond to "How did the label alone (not the calorie information or price) influence what you chose to order, if at all? The label…" with three options: more likely, less likely, or no effect
Perceived Message Effectiveness of labels | The survey will take up to 20 minutes.
  Three items averaged together:
  How much does this label discourage you from wanting to eat foods with a larger carbon footprint? [1-5: Not at all, very little, somewhat, quite a bit, a great deal]
  How much does this label make you concerned about the environmental effects of eating foods that have a larger carbon footprint? [1-5: Not at all, very little, somewhat, quite a bit, a great deal]
  How much does this label make eating foods with a larger carbon footprint seem unpleasant to you? [1-5: Not at all, very little, somewhat, quite a bit, a great deal]
Believability of labels | The survey will take up to 20 minutes.
  Item: How much do you believe this label? [1-5: Not at all, very little, somewhat, quite a bit, a great deal]
Learned from labels | The survey will take up to 20 minutes.
  Item: To what extent did you learn something new from this label? [1-5: Not at all, very little, somewhat, quite a bit, a great deal]
Talk about labels with others | The survey will take up to 20 minutes.
  Item: How likely are you to talk about this label with others? [Likert scale from not at all likely (1) to extremely likely (5)]
Understand the labels | The survey will take up to 20 minutes.
  Item: How easy or difficult was it to understand this label? [Likert scale from very easy (1) to extremely difficult (5)]

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States